CLINICAL TRIAL: NCT02639299
Title: Screening of Healthy Volunteers for Investigational Antimalarial Drugs, Malaria Vaccines, and Controlled Human Malaria Challenge
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 160039; 16-I-0039
Record Dates: First submitted 2015-12-23; First posted 2015-12-24 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12-30

CONDITIONS: Malaria
Keywords: Subjects; Venipuncture; Research; Evaluate; Recruit
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy volunteer: healthy, malaria-na(SqrRoot) ve US adults

SUMMARY:
Background:

Malaria is a serious infection caused by a parasite. People get malaria when an infected mosquito bites them. Malaria can cause major health and social problems in places were malaria is common, such as Africa but can also affect travelers who have never been exposed to malaria. Researchers at the NIH want to find a safe and effective malaria vaccine, antimalarial drugs, or prevention regimen. To do this, healthy volunteers are recruited under a general screening study in order to see if are qualified to join a future malaria study.

Objective:

To screen healthy volunteers to see if they are eligible to join investigational malaria studies. The studies will be trials of investigational antimalarial drugs, malaria vaccines, or prevention regimens. They may also involve controlled human malaria infection trials.

Eligibility:

Healthy people ages 18 50

Design:

Participants will first be prescreened by phone.

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Participants may go more than 1 year without joining a clinical trial. If this happens, they may be re-contacted to see if they still want to be part of this screening protocol. Those who still want to participate and have had relevant medical changes will be rescreened.

...

DETAILED DESCRIPTION:
This is a screening protocol for healthy volunteers to participate in research studies conducted by Laboratory of Malaria Immunology and Vaccinology (LMIV).

Malaria-related morbidity and mortality have a major economic impact in endemic regions and

present a substantial health risk to non-immune travelers and people living in endemic areas. To stem the worldwide impact of this devastating disease, a safe and broadly effective malaria vaccine and improved antimalarial therapeutics are urgently required.

This screening protocol is designed to continuously evaluate potential healthy volunteers to build a pool of volunteers who may participate in future and ongoing LMIV malaria drug, vaccine, or controlled human malaria infections (CHMI) trials. A complete medical history and blood and urine samples will be obtained to evaluate whether volunteers are eligible for study-specific screening.

ELIGIBILITY:
* INCLUSION CRITERIA:

All of the following criteria must be fulfilled for a subject to participate in this trial:

1. Age >= 18 and <= 50 years.
2. In good general health and without clinically significant medical history
3. Reliable access to the clinical trial center and available in the area for more than 1 year
4. Females of childbearing potential must be willing to undergo periodic pregnancy testing and use reliable contraception per protocol when enrolled into LMIV clinical trials (protocol-specific requirements)

EXCLUSION CRITERIA:

A subject will be excluded from participating in this trial if any one of the following criteria is fulfilled:

1. Pregnant, breastfeeding, or planned pregnancy in the upcoming year.
2. Hemoglobin, white blood cell (WBC), platelets, alanine transaminase (ALT), and creatinine (Cr) outside of local lab normal range (subjects may be included at the investigator's discretion for "not clinically significant" values outside of normal range).
3. Anticipated use during the study period, or use within the following periods prior to enrollment:

   1. Investigational malaria vaccine within the last five years
   2. Chronic systemic immunosuppressive medications (e.g., cytotoxic medications, oral/parental corticosteroids > 0.5 mg/kg/day prednisone or equivalent). Corticosteroid nasal spray for allergic rhinitis and topical corticosteroids for mild, uncomplicated dermatitis is allowed.
   3. Recurrent receipt of blood products or immunoglobulins
4. History of:

   1. Sickle cell disease
   2. Splenectomy or functional asplenia
   3. Systemic anaphylaxis
   4. Uncontrolled psoriasis or porphyria
5. Clinically significant medical condition, physical examination findings, other clinically significant abnormal laboratory results, or past medical history that may have clinically significant implications for current health status and participation in the study in the opinion of the Investigator. A clinically significant condition or process includes but is not limited to:

   1. A process that would affect the immune response, or requires medication that affects the immune response.
   2. Any contraindication to repeated phlebotomy.
6. History of or known active cardiac disease including:

   1. prior myocardial infarction (heart attack)
   2. angina pectoris
   3. congestive heart failure
   4. valvular heart disease
   5. cardiomyopathy
   6. pericarditis
   7. stroke or transient ischemic attack
   8. exertional chest pain or shortness of breath
   9. other heart conditions under the care of a doctor
7. Infection with HIV, hepatitis B, and/or hepatitis C
8. Psychiatric condition that precludes compliance with the protocol including but not limited to:

   1. Psychosis within the past 3 years
   2. Ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years
9. Suspected or known current alcohol or drug abuse as defined by the American Psychiatric Association in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition at the discretion of the PI
10. Any other finding that, in the judgment of the Investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a subject's ability to give informed consent, or increase the risk of having an adverse outcome from participating in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers in the Washington, DC region
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-12-08 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
To screen healthy volunteers for future malaria studies | 1 year
  identify healthy adults at a low risk of developing complications due to experimental malaria infection, investigational antimalarials and vaccines

CONTACTS AND LOCATIONS:
Overall Officials: David M Cook, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
This is a screening protocol for healthy volunteers to participate in research studies conducted by Laboratory of Malaria Immunology and Vaccinology (LMIV).@@@@@@@@@@@@This screening protocol is designed to evaluate potential healthy volunteers to build a pool of volunteers who may participate in future and ongoing LMIV malaria drug, vaccine, or controlled human malaria infections (CHMI) trials. Data obtained for individual subjects will used not be used for direct research purposes on this study; therefore we will not make IPD available at this time.

REFERENCES:
- [Background] YOELI M. STUDIES ON PLASMODIUM BERGHEI IN NATURE AND UNDER EXPERIMENTAL CONDITIONS. Trans R Soc Trop Med Hyg. 1965 May;59:255-76. doi: 10.1016/0035-9203(65)90004-0. No abstract available. PMID 14298028
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2016-I-0039.html